CLINICAL TRIAL: NCT05487885
Title: Anhedonia, Development, and Emotions: Phenotyping and Therapeutics (ADEPT) Study
Brief Title: Anhedonia, Development, and Emotions: Phenotyping and Therapeutics
Acronym: ADEPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erika Forbes (Other)
Responsible Party: Sponsor-Investigator, Erika Forbes, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21120080
Record Dates: First submitted 2022-07-27; First posted 2022-08-04 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Depression; Anhedonia
Keywords: depression; anhedonia
MeSH Terms: conditions — Depression; Anhedonia

STUDY DESIGN:
Intervention Model Description: The study has a longitudinal design in which participants complete 2 sets of activities:
  Phase 1: Phenotyping. This includes assessment with diagnostic interview, questionnaires, behavioral tasks, MRI, app-based digital assessment, and blood draw for inflammatory markers. This set of activities will occur at 4 time points over the course of 1 year/participant (study entry, approximately 4 months, approximately 5 months, and approximately 1 year), and all participants will complete them.
  Phase 2: Therapeutic activities: (1) 10 theta burst stimulation (TBS) sessions (TBS 2 times/session) plus positive affect (PA) training for all participants; and (2) IV ketamine infusion for those who do not respond to TBS/PA activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TMS and PAT (Experimental): All open label with no randomization to placebo
  Interventions: Device: Continuous theta burst stimulation (cTBS); Behavioral: Positive Affect Training
- TMS and PAT, then Ketamine (Experimental): All open label with no randomization to placebo
  Interventions: Device: Continuous theta burst stimulation (cTBS); Behavioral: Positive Affect Training; Drug: Ketamine Injectable Solution

INTERVENTIONS:
Device: Continuous theta burst stimulation (cTBS) — a form of transcranial magnetic stimulation, to dorsomedial prefrontal cortex (dmPFC)
Behavioral: Positive Affect Training — Psychosocial add-on intervention that could enhance the effects of TBS. PA Therapy (Craske et al., 2016) is an innovative cognitive and experiential technique developed to address anhedonia specifically and, ideally, change altered patterns of frontostriatal function. Standing in contrast to Cognitive Behavioral Therapy, PA training has efficacy for enhancing positive affect and reducing negative affect (Craske et al., 2018). This treatment can be easily applied, and we propose that it will enhance neural circuit-level changes elicited by TBS.
Drug: Ketamine Injectable Solution — Ketamine is FDA-approved as an anesthetic agent that will be used off-label in this study. It is used routinely in both pediatric and adult patients and is considered extremely safe in substantially higher, anesthetic doses. The dose to be administered here (0.5 mg/kg) is a much lower, subanesthetic dose, and the administration route (intravenous) is the standard when used in anesthesia. Published studies and metaanalyses of this dose of intravenous ketamine as an off label use in depression show clearly that there are no increased risks in this population, including a recent study in adolescents (Dwyer et al, 2021, American Journal of Psychiatry). A single dose of ketamine will be used to determine if it alters the functioning of the anhedonia-related reward functioning and frontostriatal biomarkers assessed in this study.
  Arms: TMS and PAT, then Ketamine

SUMMARY:
The goal of the ADEPT Study is to understand anhedonia in young people and how it changes based on treatments targeting the brain circuit underlying it. Anhedonia is a challenging mental health symptom that involves difficulty with motivation to experience pleasant events. This study could help develop treatments for people whose depression does not improve with traditional treatments.

The ADEPT Study includes two phases. In Phase 1, participants are asked to go through a series of activities to measure anhedonia, including MRI scans, blood draws, behavioral tasks, clinical interviews, questionnaires, and app-based assessments of experiences and behaviors. Phase 2 involves therapeutic activities, such as transcranial magnetic stimulation (TMS), positive affect training, and, for some people, ketamine administration. If the participant qualifies and is interested, they may choose to do Phase 2 activities in addition to Phase 1.

DETAILED DESCRIPTION:
In this research study, the investigators are trying to understand and change anhedonia in young people with depression. Anhedonia is experienced by many people who have depression, and it involves difficulty with motivation, energy, and anticipation of pleasant events. People who experience anhedonia often have more severe depression, experience depression for longer periods of time, and don't easily get better with traditional treatments. The investigators want to understand anhedonia early in life in order to help young people develop along healthy pathways and avoid chronic illness. Anhedonia is related to function in the brain's reward circuit, inflammation in the body, and people's experiences and behaviors, and will measure all of these. The investigators also want to understand anhedonia by using treatments that could improve it. To do that, activities will be used that have been used to treat depression and target the brain's reward circuit, which is believed to be the source of anhedonia. Finally, anhedonia will be measured over approximately 1 year to see how it changes with time, development, or treatment-based experiences. Eventually, the findings of this study might be useful for treating depression and improving people's quality of life.

The study is looking for 300 young people (aged 15-25) who are currently experiencing depression to participate in our research study. In Phase 1 of our study, a series of activities will be conducted to understand the characteristics of anhedonia, including MRI scans, blood draws, behavioral tasks, clinical interviews, questionnaires, and measurement of real-life experiences and behavior using a phone app. This is called "phenotyping" because these characteristics are also called phenotypes.

The eligibility process for Phase 1 will include an interview with questions about the participant's mood, experiences, and behaviors. This interview will take approximately 2-3 hours. With permission, interviews will be video recorded to facilitate training and supervision of study staff. Participants will also be asked questions about health, including treatment history.

Study procedures include 4 visits over approximately 1 year. These may be broken into two sessions per visit for scheduling reasons. In addition, the study will include an ongoing smartphone app-based assessment of mood, experiences, and behavior.

Visit 1 consists of an MRI scan, questionnaires about thoughts, emotions, and experiences, tasks on a computer and a blood draw by a trained phlebotomist. Visits 2-4 consists of a second MRI scan, questionnaires, tasks on a computer, a blood draw by a trained phlebotomist, and an interview about mood, experiences, and behaviors.

Phase 2 of this study involves procedures that are therapeutic, meaning they can treat depression and anhedonia. These include transcranial magnetic stimulation (TMS), which is a noninvasive procedure to treat depression that uses magnetic fields to stimulate nerve cells in the brain. Visits with TMS will include Positive Affect Training, which involves changing behaviors and thoughts to build positive emotions. People whose depression does not improve with TMS may receive a single intravenous (IV, or into the vein) infusion of ketamine, a medicine that is used in hospitals for anesthesia and that can improve depression quickly.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 (all participants)

* Current DSM-5 depressive disorder
* Severity ≥ 12 on MADRS
* Moderate-severe anhedonia (75% of sample) or low anhedonia (25% of sample)

Phase 2 (for participants in TBS and ketamine phase, in addition to above)

• ≥ 1 failed antidepressant trial (for qualification for Phase 2 of study and definition of non-response to TMS in order to be eligible for ketamine) = Treatment for at least 6 weeks with an antidepressant medication reaching recommended dosage for adults for at least 3 weeks of the treatment (e.g., 20 mg fluoxetine)

Exclusion Criteria:

Phase 1 (all participants)

* Lifetime psychosis, bipolar disorder, or developmental disorder
* Serious, unstable neurological disorder (e.g., seizure disorder)
* Brain injury with loss of consciousness
* Moderate-severe substance use disorder, past 6 mos.
* MRI contraindications (e.g., metal in body)

Phase 2 (for participants in TBS and ketamine phase, in addition to above)

* Serious, unstable respiratory or cardiovascular illness
* Pre-TBS: Alcohol binge in past week or > 3 drinks/day in past 3 days
* Pre-ketamine: use of MAOIs in past 2 weeks
* Pregnancy
* High blood pressure
* Current illicit stimulant use
* Lifetime recreational ketamine or PCP use

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) score | pre- to post-TMS (over 2 weeks)
  This clinician-rated scale captures depression severity on a scale of 0-60, with higher scores reflecting greater severity

SECONDARY OUTCOMES:
Snaith Hamilton Pleasure Scale (SHAPS) score | pre- to post-TMS (over 2 weeks)
  This 14-item self-report questionnaire measures anhedonia, or difficulty with motivation toward or enjoyment of pleasant events. Total scores range from 14-56, with higher scores reflecting greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Erika E Forbes, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Loeffler Building, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aquino D, Bizzi A, Grisoli M, Garavaglia B, Bruzzone MG, Nardocci N, Savoiardo M, Chiapparini L. Age-related iron deposition in the basal ganglia: quantitative analysis in healthy subjects. Radiology. 2009 Jul;252(1):165-72. doi: 10.1148/radiol.2522081399. PMID 19561255
- [Background] Belujon P, Grace AA. Dopamine System Dysregulation in Major Depressive Disorders. Int J Neuropsychopharmacol. 2017 Dec 1;20(12):1036-1046. doi: 10.1093/ijnp/pyx056. PMID 29106542
- [Background] Berridge KC. Evolving Concepts of Emotion and Motivation. Front Psychol. 2018 Sep 7;9:1647. doi: 10.3389/fpsyg.2018.01647. eCollection 2018. PMID 30245654
- [Background] Boyle CC, Kuhlman KR, Dooley LN, Haydon MD, Robles TF, Ang YS, Pizzagalli DA, Bower JE. Inflammation and dimensions of reward processing following exposure to the influenza vaccine. Psychoneuroendocrinology. 2019 Apr;102:16-23. doi: 10.1016/j.psyneuen.2018.11.024. Epub 2018 Nov 20. PMID 30496908
- [Background] Brenhouse HC, Schwarz JM. Immunoadolescence: Neuroimmune development and adolescent behavior. Neurosci Biobehav Rev. 2016 Nov;70:288-299. doi: 10.1016/j.neubiorev.2016.05.035. Epub 2016 May 31. PMID 27260127
- [Background] Brundin L, Bryleva EY, Thirtamara Rajamani K. Role of Inflammation in Suicide: From Mechanisms to Treatment. Neuropsychopharmacology. 2017 Jan;42(1):271-283. doi: 10.1038/npp.2016.116. Epub 2016 Jul 5. PMID 27377015
- [Background] Cassidy CM, Zucca FA, Girgis RR, Baker SC, Weinstein JJ, Sharp ME, Bellei C, Valmadre A, Vanegas N, Kegeles LS, Brucato G, Kang UJ, Sulzer D, Zecca L, Abi-Dargham A, Horga G. Neuromelanin-sensitive MRI as a noninvasive proxy measure of dopamine function in the human brain. Proc Natl Acad Sci U S A. 2019 Mar 12;116(11):5108-5117. doi: 10.1073/pnas.1807983116. Epub 2019 Feb 22. PMID 30796187
- [Background] Chase HW, Fournier JC, Bertocci MA, Greenberg T, Aslam H, Stiffler R, Lockovich J, Graur S, Bebko G, Forbes EE, Phillips ML. A pathway linking reward circuitry, impulsive sensation-seeking and risky decision-making in young adults: identifying neural markers for new interventions. Transl Psychiatry. 2017 Apr 18;7(4):e1096. doi: 10.1038/tp.2017.60. PMID 28418404
- [Background] Chen X, Huddleston DE, Langley J, Ahn S, Barnum CJ, Factor SA, Levey AI, Hu X. Simultaneous imaging of locus coeruleus and substantia nigra with a quantitative neuromelanin MRI approach. Magn Reson Imaging. 2014 Dec;32(10):1301-6. doi: 10.1016/j.mri.2014.07.003. Epub 2014 Jul 31. PMID 25086330
- [Background] Connor JR, Menzies SL. Relationship of iron to oligodendrocytes and myelination. Glia. 1996 Jun;17(2):83-93. doi: 10.1002/(SICI)1098-1136(199606)17:23.0.CO;2-7. PMID 8776576
- [Background] Cosgrove KT, Burrows K, Avery JA, Kerr KL, DeVille DC, Aupperle RL, Teague TK, Drevets WC, Simmons WK. Appetite change profiles in depression exhibit differential relationships between systemic inflammation and activity in reward and interoceptive neurocircuitry. Brain Behav Immun. 2020 Jan;83:163-171. doi: 10.1016/j.bbi.2019.10.006. Epub 2019 Oct 8. PMID 31604141
- [Background] Craske MG, Meuret AE, Ritz T, Treanor M, Dour HJ. Treatment for Anhedonia: A Neuroscience Driven Approach. Depress Anxiety. 2016 Oct;33(10):927-938. doi: 10.1002/da.22490. PMID 27699943
- [Background] Craske MG, Meuret AE, Ritz T, Treanor M, Dour H, Rosenfield D. Positive affect treatment for depression and anxiety: A randomized clinical trial for a core feature of anhedonia. J Consult Clin Psychol. 2019 May;87(5):457-471. doi: 10.1037/ccp0000396. PMID 30998048
- [Background] Der-Avakian A, Barnes SA, Markou A, Pizzagalli DA. Translational Assessment of Reward and Motivational Deficits in Psychiatric Disorders. Curr Top Behav Neurosci. 2016;28:231-62. doi: 10.1007/7854_2015_5004. PMID 26873017
- [Background] Der-Avakian A, Markou A. The neurobiology of anhedonia and other reward-related deficits. Trends Neurosci. 2012 Jan;35(1):68-77. doi: 10.1016/j.tins.2011.11.005. Epub 2011 Dec 15. PMID 22177980
- [Background] Drysdale AT, Grosenick L, Downar J, Dunlop K, Mansouri F, Meng Y, Fetcho RN, Zebley B, Oathes DJ, Etkin A, Schatzberg AF, Sudheimer K, Keller J, Mayberg HS, Gunning FM, Alexopoulos GS, Fox MD, Pascual-Leone A, Voss HU, Casey BJ, Dubin MJ, Liston C. Resting-state connectivity biomarkers define neurophysiological subtypes of depression. Nat Med. 2017 Jan;23(1):28-38. doi: 10.1038/nm.4246. Epub 2016 Dec 5. PMID 27918562
- [Background] Dwyer JB, Landeros-Weisenberger A, Johnson JA, Londono Tobon A, Flores JM, Nasir M, Couloures K, Sanacora G, Bloch MH. Efficacy of Intravenous Ketamine in Adolescent Treatment-Resistant Depression: A Randomized Midazolam-Controlled Trial. Am J Psychiatry. 2021 Apr 1;178(4):352-362. doi: 10.1176/appi.ajp.2020.20010018. Epub 2021 Mar 3. PMID 33653121
- [Background] Felger JC. The Role of Dopamine in Inflammation-Associated Depression: Mechanisms and Therapeutic Implications. Curr Top Behav Neurosci. 2017;31:199-219. doi: 10.1007/7854_2016_13. PMID 27225499
- [Background] Felger JC, Li Z, Haroon E, Woolwine BJ, Jung MY, Hu X, Miller AH. Inflammation is associated with decreased functional connectivity within corticostriatal reward circuitry in depression. Mol Psychiatry. 2016 Oct;21(10):1358-65. doi: 10.1038/mp.2015.168. Epub 2015 Nov 10. PMID 26552591
- [Background] Felger JC, Treadway MT. Inflammation Effects on Motivation and Motor Activity: Role of Dopamine. Neuropsychopharmacology. 2017 Jan;42(1):216-241. doi: 10.1038/npp.2016.143. Epub 2016 Aug 2. PMID 27480574
- [Background] Forbes EE, Dahl RE. Research Review: altered reward function in adolescent depression: what, when and how? J Child Psychol Psychiatry. 2012 Jan;53(1):3-15. doi: 10.1111/j.1469-7610.2011.02477.x. Epub 2011 Nov 28. PMID 22117893
- [Background] Forbes EE, Hariri AR, Martin SL, Silk JS, Moyles DL, Fisher PM, Brown SM, Ryan ND, Birmaher B, Axelson DA, Dahl RE. Altered striatal activation predicting real-world positive affect in adolescent major depressive disorder. Am J Psychiatry. 2009 Jan;166(1):64-73. doi: 10.1176/appi.ajp.2008.07081336. Epub 2008 Dec 1. PMID 19047324
- [Background] Friedman J, Hastie T, Tibshirani R. glmnet: Lasso and elastic-net regularized generalized linear models. Version1. 2013.
- [Background] Goldsworthy MR, Rogasch NC, Ballinger S, Graetz L, Van Dam JM, Harris R, Yu S, Pitcher JB, Baune BT, Ridding MC. Age-related decline of neuroplasticity to intermittent theta burst stimulation of the lateral prefrontal cortex and its relationship with late-life memory performance. Clin Neurophysiol. 2020 Sep;131(9):2181-2191. doi: 10.1016/j.clinph.2020.06.015. Epub 2020 Jul 3. PMID 32693192
- [Background] Haacke EM, Cheng NY, House MJ, Liu Q, Neelavalli J, Ogg RJ, Khan A, Ayaz M, Kirsch W, Obenaus A. Imaging iron stores in the brain using magnetic resonance imaging. Magn Reson Imaging. 2005 Jan;23(1):1-25. doi: 10.1016/j.mri.2004.10.001. PMID 15733784
- [Background] Healey KL, Morgan J, Musselman SC, Olino TM, Forbes EE. Social anhedonia and medial prefrontal response to mutual liking in late adolescents. Brain Cogn. 2014 Aug;89:39-50. doi: 10.1016/j.bandc.2013.12.004. Epub 2014 Jan 10. PMID 24412087
- [Background] Hordacre B, Goldsworthy MR, Graetz L, Ridding MC. Motor network connectivity predicts neuroplastic response following theta burst stimulation in healthy adults. Brain Struct Funct. 2021 Jul;226(6):1893-1907. doi: 10.1007/s00429-021-02299-4. Epub 2021 May 27. PMID 34043076
- [Background] Jones BDM, Daskalakis ZJ, Carvalho AF, Strawbridge R, Young AH, Mulsant BH, Husain MI. Inflammation as a treatment target in mood disorders: review. BJPsych Open. 2020 Jun 5;6(4):e60. doi: 10.1192/bjo.2020.43. PMID 32498754
- [Background] Keren H, O'Callaghan G, Vidal-Ribas P, Buzzell GA, Brotman MA, Leibenluft E, Pan PM, Meffert L, Kaiser A, Wolke S, Pine DS, Stringaris A. Reward Processing in Depression: A Conceptual and Meta-Analytic Review Across fMRI and EEG Studies. Am J Psychiatry. 2018 Nov 1;175(11):1111-1120. doi: 10.1176/appi.ajp.2018.17101124. Epub 2018 Jun 20. PMID 29921146
- [Background] Kuhlman KR, Chiang JJ, Horn S, Bower JE. Developmental psychoneuroendocrine and psychoneuroimmune pathways from childhood adversity to disease. Neurosci Biobehav Rev. 2017 Sep;80:166-184. doi: 10.1016/j.neubiorev.2017.05.020. Epub 2017 May 31. PMID 28577879
- [Background] Larsen B, Luna B. In vivo evidence of neurophysiological maturation of the human adolescent striatum. Dev Cogn Neurosci. 2015 Apr;12:74-85. doi: 10.1016/j.dcn.2014.12.003. Epub 2014 Dec 30. PMID 25594607
- [Background] Lally N, Nugent AC, Luckenbaugh DA, Ameli R, Roiser JP, Zarate CA. Anti-anhedonic effect of ketamine and its neural correlates in treatment-resistant bipolar depression. Transl Psychiatry. 2014 Oct 14;4(10):e469. doi: 10.1038/tp.2014.105. PMID 25313512
- [Background] Lally N, Nugent AC, Luckenbaugh DA, Niciu MJ, Roiser JP, Zarate CA Jr. Neural correlates of change in major depressive disorder anhedonia following open-label ketamine. J Psychopharmacol. 2015 May;29(5):596-607. doi: 10.1177/0269881114568041. Epub 2015 Feb 17. PMID 25691504
- [Background] Larsen B, Olafsson V, Calabro F, Laymon C, Tervo-Clemmens B, Campbell E, Minhas D, Montez D, Price J, Luna B. Maturation of the human striatal dopamine system revealed by PET and quantitative MRI. Nat Commun. 2020 Feb 12;11(1):846. doi: 10.1038/s41467-020-14693-3. PMID 32051403
- [Background] Lin A, Yung AR, Wigman JT, Killackey E, Baksheev G, Wardenaar KJ. Validation of a short adaptation of the Mood and Anxiety Symptoms Questionnaire (MASQ) in adolescents and young adults. Psychiatry Res. 2014 Mar 30;215(3):778-83. doi: 10.1016/j.psychres.2013.12.018. Epub 2013 Dec 18. PMID 24387880
- [Background] McMakin DL, Olino TM, Porta G, Dietz LJ, Emslie G, Clarke G, Wagner KD, Asarnow JR, Ryan ND, Birmaher B, Shamseddeen W, Mayes T, Kennard B, Spirito A, Keller M, Lynch FL, Dickerson JF, Brent DA. Anhedonia predicts poorer recovery among youth with selective serotonin reuptake inhibitor treatment-resistant depression. J Am Acad Child Adolesc Psychiatry. 2012 Apr;51(4):404-11. doi: 10.1016/j.jaac.2012.01.011. Epub 2012 Mar 3. PMID 22449646
- [Background] Miller AH, Raison CL. The role of inflammation in depression: from evolutionary imperative to modern treatment target. Nat Rev Immunol. 2016 Jan;16(1):22-34. doi: 10.1038/nri.2015.5. PMID 26711676
- [Background] Mitchell RH, Goldstein BI. Inflammation in children and adolescents with neuropsychiatric disorders: a systematic review. J Am Acad Child Adolesc Psychiatry. 2014 Mar;53(3):274-96. doi: 10.1016/j.jaac.2013.11.013. Epub 2013 Dec 16. PMID 24565356
- [Background] Moeini M, Khaleghi A, Mohammadi MR. Characteristics of Alpha Band Frequency in Adolescents with Bipolar II Disorder: A Resting-State QEEG Study. Iran J Psychiatry. 2015;10(1):8-12. PMID 26005474
- [Background] Nance M, Eckstrand KL, Lindenmuth M, Ambrosia M, Forbes EE. Adolescents' medial prefrontal cortex response to monetary reward mediates the association between C-reactive protein and anhedonia 6 months later. In preparation.
- [Background] Ortega R, Cloetens P, Deves G, Carmona A, Bohic S. Iron storage within dopamine neurovesicles revealed by chemical nano-imaging. PLoS One. 2007 Sep 26;2(9):e925. doi: 10.1371/journal.pone.0000925. PMID 17895967
- [Background] Osugi Y, Hara J, Kurahashi H, Sakata N, Inoue M, Yumura-Yagi K, Kawa-Ha K, Okada S, Tawa A. Age-related changes in surface antigens on peripheral lymphocytes of healthy children. Clin Exp Immunol. 1995 Jun;100(3):543-8. doi: 10.1111/j.1365-2249.1995.tb03735.x. PMID 7774067
- [Background] Parr AC, Calabro F, Larsen B, Tervo-Clemmens B, Elliot S, Foran W, Olafsson V, Luna B. Dopamine-related striatal neurophysiology is associated with specialization of frontostriatal reward circuitry through adolescence. Prog Neurobiol. 2021 Jun;201:101997. doi: 10.1016/j.pneurobio.2021.101997. Epub 2021 Mar 2. PMID 33667595
- [Background] Pizzagalli DA. Depression, stress, and anhedonia: toward a synthesis and integrated model. Annu Rev Clin Psychol. 2014;10:393-423. doi: 10.1146/annurev-clinpsy-050212-185606. PMID 24471371
- [Background] Pratt LA, Brody DJ, Gu Q. Antidepressant use in persons aged 12 and over: United States, 2005-2008. NCHS Data Brief. 2011 Oct;(76):1-8. PMID 22617183
- [Background] Pulcu E, Guinea C, Cowen PJ, Murphy SE, Harmer CJ. A translational perspective on the anti-anhedonic effect of ketamine and its neural underpinnings. Mol Psychiatry. 2022 Jan;27(1):81-87. doi: 10.1038/s41380-021-01183-1. Epub 2021 Jun 22. PMID 34158619
- [Background] Radloff LS. The CES-D scale: A self-report depression scale for research in the general population. Applied psychological measurement. 1977;1(3):385-401.
- [Background] Rajapakse T, Kirton A. NON-INVASIVE BRAIN STIMULATION IN CHILDREN: APPLICATIONS AND FUTURE DIRECTIONS. Transl Neurosci. 2013 Jun;4(2):10.2478/s13380-013-0116-3. doi: 10.2478/s13380-013-0116-3. PMID 24163755
- [Background] Rizvi SJ, Pizzagalli DA, Sproule BA, Kennedy SH. Assessing anhedonia in depression: Potentials and pitfalls. Neurosci Biobehav Rev. 2016 Jun;65:21-35. doi: 10.1016/j.neubiorev.2016.03.004. Epub 2016 Mar 6. PMID 26959336
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Somerville LH, Casey BJ. Developmental neurobiology of cognitive control and motivational systems. Curr Opin Neurobiol. 2010 Apr;20(2):236-41. doi: 10.1016/j.conb.2010.01.006. Epub 2010 Feb 16. PMID 20167473
- [Background] Sulzer D, Cassidy C, Horga G, Kang UJ, Fahn S, Casella L, Pezzoli G, Langley J, Hu XP, Zucca FA, Isaias IU, Zecca L. Neuromelanin detection by magnetic resonance imaging (MRI) and its promise as a biomarker for Parkinson's disease. NPJ Parkinsons Dis. 2018 Apr 10;4:11. doi: 10.1038/s41531-018-0047-3. eCollection 2018. PMID 29644335
- [Background] Treadway MT, Buckholtz JW, Schwartzman AN, Lambert WE, Zald DH. Worth the 'EEfRT'? The effort expenditure for rewards task as an objective measure of motivation and anhedonia. PLoS One. 2009 Aug 12;4(8):e6598. doi: 10.1371/journal.pone.0006598. PMID 19672310
- [Background] Treadway MT, Zald DH. Reconsidering anhedonia in depression: lessons from translational neuroscience. Neurosci Biobehav Rev. 2011 Jan;35(3):537-55. doi: 10.1016/j.neubiorev.2010.06.006. Epub 2010 Jul 11. PMID 20603146
- [Background] Wang Y, Butros SR, Shuai X, Dai Y, Chen C, Liu M, Haacke EM, Hu J, Xu H. Different iron-deposition patterns of multiple system atrophy with predominant parkinsonism and idiopathetic Parkinson diseases demonstrated by phase-corrected susceptibility-weighted imaging. AJNR Am J Neuroradiol. 2012 Feb;33(2):266-73. doi: 10.3174/ajnr.A2765. Epub 2011 Nov 3. PMID 22051807
- [Background] Wang L, Li F, Mitchell PB, Wang CY, Si TM. Striatal Resting-State Connectivity Abnormalities Associated With Different Clinical Stages of Major Depressive Disorder. J Clin Psychiatry. 2020 Feb 18;81(2):19m12790. doi: 10.4088/JCP.19m12790. PMID 32078260
- [Background] Ward RJ, Zucca FA, Duyn JH, Crichton RR, Zecca L. The role of iron in brain ageing and neurodegenerative disorders. Lancet Neurol. 2014 Oct;13(10):1045-60. doi: 10.1016/S1474-4422(14)70117-6. PMID 25231526
- [Background] Wengler K, He X, Abi-Dargham A, Horga G. Reproducibility assessment of neuromelanin-sensitive magnetic resonance imaging protocols for region-of-interest and voxelwise analyses. Neuroimage. 2020 Mar;208:116457. doi: 10.1016/j.neuroimage.2019.116457. Epub 2019 Dec 11. PMID 31841683
- [Background] Whitton AE, Treadway MT, Pizzagalli DA. Reward processing dysfunction in major depression, bipolar disorder and schizophrenia. Curr Opin Psychiatry. 2015 Jan;28(1):7-12. doi: 10.1097/YCO.0000000000000122. PMID 25415499
- [Background] Xing Y, Sapuan A, Dineen RA, Auer DP. Life span pigmentation changes of the substantia nigra detected by neuromelanin-sensitive MRI. Mov Disord. 2018 Nov;33(11):1792-1799. doi: 10.1002/mds.27502. Epub 2018 Nov 13. PMID 30423212
- [Background] Zhang WN, Chang SH, Guo LY, Zhang KL, Wang J. The neural correlates of reward-related processing in major depressive disorder: a meta-analysis of functional magnetic resonance imaging studies. J Affect Disord. 2013 Nov;151(2):531-539. doi: 10.1016/j.jad.2013.06.039. Epub 2013 Jul 12. PMID 23856280
- [Background] Zucca FA, Segura-Aguilar J, Ferrari E, Munoz P, Paris I, Sulzer D, Sarna T, Casella L, Zecca L. Interactions of iron, dopamine and neuromelanin pathways in brain aging and Parkinson's disease. Prog Neurobiol. 2017 Aug;155:96-119. doi: 10.1016/j.pneurobio.2015.09.012. Epub 2015 Oct 9. PMID 26455458